CLINICAL TRIAL: NCT01361321
Title: Examining Bone Quantity and Quality Following Standard Guided Bone Regeneration Procedures
Brief Title: Bone Quality and Quantity Following Guided Bone Regeneration
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: bondbone-HMO-CTIL
Record Dates: First submitted 2011-05-18; First posted 2011-05-26 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2013-09

CONDITIONS: Alveolar Ridge Augmentation
Keywords: follow up; Guided bone regeneration; Micro computerized tomography; histological examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Reisdual bone tissue formed while preparing alveolar bone for dental implant (by drilling with a trephine bur)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients after GBR procedure: The study will comprise of patients who already underwent a routine Guided Bone Regeneration (GBR) procedure in order to augment a bony ridge before dental implant insertion. The patients will be followed up in order to determine bone quality and quantity formed after the usage of routinely used bone substitutes during GBR procedure.

SUMMARY:
Edentulism refers to a state of full or partial lack of teeth. This situation may interfere with essential functions such as mastication, speech and even appearance.

Dental implants inserted to the mandible or maxilla is a common treatment modality aiming to restore edentulus alveolar ridges by providing support and anchorage for removable or fixed dental prosthesis.There are cases which in addition to a lack of teeth suffer from lack of sufficient bone tissue volume to support the dental implant.A situation like this may originate from a variety of reasons such as residual bone atrophy, prior alveolar bone destruction due to periodontal disease and even a traumatic tooth extraction. In such cases, a routine alveolar bone augmentation is done to enable a dental implant installation at this site.Guided bone regeneration (GBR) is a widely used technique used to augment edentulus bone ridges. It relies on an inert membrane covering a bone substitute placed over the bony site requiring augmentation. The bone substitute provides a scaffold to alveolar regeneration by the host's osteoblasts while the membrane prevents unwanted epithelial cells to migrate to the bony defect area.

The investigators research is a aimed to preform a follow up after patients who already went through a GBR procedure and before inserting a dental implant. Patients answering the inclusion but not the exclusion criteria will go through an alveolar computerized tomography (C.T) done routinely before inserting dental implants.At the day of Dental implantation - residual bone left from the site of implantation (after preparing the site with a trephine bur) will be taken to a histological analysis. The results from the C.T and the histological examination will be analyzed for bone quantity (volume) and quality and will allow a comparison of bone characteristics obtained by using different routinely used bone substitutes.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women over 18 years of age, eligible for signing
2. Patients who went through a GBR procedure previous to an insertion of a dental implant which hasn't been inserted yet
3. Patients who understand the meaning of the treatment (routine dental implant insertion) and the follow up study, and approves participation in booth of them

Exclusion Criteria:

1. Pregnant or nursing women. children or non judgemental patients
2. Patients with uncontrolled diabetas mellitus, rheumatoid arthritis or osteoporosis.
3. Patients with a pathology present near the site of dental implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healty over 18 years of age Patients who went through a GBR procedure previous to an insertion of a dental implant which hasn't been insertd yet
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02-21 (Actual); Study Completion 2013-02-21 (Actual)

PRIMARY OUTCOMES:
Volume of the new bone formed after a GBR procedure | Volume of the new bone formed after the GBR procedure will be determined 6-7 months after the GBR procedure and before the insertion of dental implants.
  Bone volume obtained following a GBR procedure will be detemined through a comparison of a 3 dimensional analysis of computed tomography images done before and after the GBR procedure.

SECONDARY OUTCOMES:
Bone quality | Bone quality will be assesed through histological analysis that will be carried out at the time of implants insertion 7-8 months after the GBR procedure.
  The collected bone sample will be subjected to histo-morphometric analysis in order to determine the size, shape and orientation of the bony trabeculae,the size and porosity of the bony cortex in addition to the new bone/ bone substitute ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Shapira, Professor, Principal Investigator — Department of Periodontology
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel